CLINICAL TRIAL: NCT02840058
Title: Interest of Anti-telomerase T CD4 Immune Responses for Predicting the Effectiveness of Immunotherapies Targeting PD1 / PDL1
Acronym: ITHER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: API/2015/58
Record Dates: First submitted 2016-07-13; First posted 2016-07-21 (Estimated); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Biological samples (Experimental): Blood samples will be realized specifically to the study at inclusion (baseline before starting anti PD1/PDL1 treatment), and then 1 month, 3 months and 12 months after initiation of anti-PD1/PDL1 treatment.
  Peripheral blood mononuclear cells (PBMC) and plasma will be collected.
  Available tumor tissues will be collected.
  Interventions: Other: Biological samples; Drug: Anti PD1/PDL1 treatment

INTERVENTIONS:
Other: Biological samples — blood and tumor tissue samples
Drug: Anti PD1/PDL1 treatment

SUMMARY:
Recent scientific advances have shown the important role of immune system against cancer. Today, many immunological biotherapy like anti-PD1/PDL-1 are available in cancer treatment and generate durable clinical responses in some patients. The development of tools for monitoring anti-tumor immune responses dynamically is a major challenge to predict the effectiveness of immunotherapies anti-PD-1 and anti-PDL-1.

Thus, the objective of our study is to analyse the interest of the monitoring of anti-telomerase T helper 1 (TH1) responses in predicting the efficacy of immunotherapy, using an immunoassay developed by our group.

ELIGIBILITY:
Inclusion Criteria:

* Patient with metastatic or locally advanced cancer candidate to anti-PD1/PDL1 immunotherapy
* Performance status 0, 1 or 2 on the ECOG scale
* Written informed consent

Exclusion Criteria:

* Patients under chronic treatment with systemic corticoids or other immunosuppressive drugs (prednisone or prednisolone ≤ 10 mg/day is allowed)
* Prior history of other malignancy except for: basal cell carcinoma of the skin, cervical intra-epithelial neoplasia and other cancer curatively treated with no evidence of disease for at least 5 years
* Active autoimmune diseases, HIV, hepatitis C or B virus
* Patients with any medical or psychiatric condition or disease,
* Patients under guardianship, curatorship or under the protection of justice.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-07 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
anti-telomerase specific Th1 responses | up to 12 months after the initiation of anti-PD1/PDL1 therapy
  measured by ELISPOT assay
objective response rate | up to 12 months after the initiation of anti-PD1/PDL1 therapy
  according to RECIST v1.1 criteria

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Besançon, Besançon, France